CLINICAL TRIAL: NCT04160780
Title: Lateral Sinus Augmentation Using L-PRF and Xenograft: Radiographic and Histomorphometry Analysis.
Brief Title: Lateral Sinus Augmentation Using L-PRF as Sole Graft Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Alhassan Diab, assistant lecturer, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 280986
Record Dates: First submitted 2019-09-08; First posted 2019-11-13 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Maxillary Diseases
MeSH Terms: conditions — Maxillary Diseases | interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-PRF as sole graft material (Experimental): lateral sinus augmentation using L-PRF as sole graft material
  Interventions: Procedure: L-PRF
- xenograft as sole graft material (Experimental): lateral sinus augmentation using xenograft as sole graft material
  Interventions: Procedure: xenograft
- Xenograft mixed with L-PRF as graft material (Experimental): lateral sinus augmentation using L-PRF mixed with xenograft as graft material
  Interventions: Procedure: L-PRF mixed with xenograft

INTERVENTIONS:
Procedure: L-PRF — sinus augmentation using L-PRf as sole graft material
  Arms: L-PRF as sole graft material
Procedure: L-PRF mixed with xenograft — sinus augmentation using L-PRF mixed with xenograft as sole graft material
  Arms: Xenograft mixed with L-PRF as graft material
Procedure: xenograft — sinus augmentation using xenograft as sole graft material
  Arms: xenograft as sole graft material

SUMMARY:
Severe maxillary atrophy occurs after extraction of teeth in poster maxilla due to dimensional changes occur after removal; besides, sinus membrane pneumatization causes alveolar bone resorption, different classification for remaining alveolar bone in the posterior maxilla were done. In this study, the ABC sinus classification was followed in case selection. A sinus augmentation is done with several techniques. Sinus membrane elevation is done with two different approaches, either the crestal approach or lateral window approach.

Using biofiller material for sinus membrane elevation has been tried by many researchers, using a bone graft, platelet concentrates preparation, collagen membranes, tenting screws, or with implant tenting.

In this study, sinus augmentation was performed using a lateral window approach using L-PRF as sole biofiller material in one group, xenograft as only biofiller material in the second group and mixed xenograft with L-PRF in the third group. Histomorphometric analysis was done from the core biopsy after three months of augmentation, and implant placement was done.

After three months, prosthetic parts were placed. The results of this study show that the augmentation of the sinus using L-PRF mixed with bone graft is showing the best results followed by L-PRF only, and the least was xenograft.

From this point of discussion, it can be considered that using L-PRF as sole biofiller material in sinus augmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult patients.
2. Both sex, males and females.
3. Age from 24 - 49 years old.
4. All patients were free from any systemic diseases as evidenced by Burkett's oral medicine health history questionnaire.
5. Extraction done at posterior maxilla involved with the maxillary sinus.
6. Remaining alveolar bone ≤ 5mm vertically and ≥ 4mm horizontally and from 1.5 mm to 3.5 mm vertically.
7. Gingival biotype 1-2mm thickness.
8. Patient has no previous surgery in Maxillary antrum.

Exclusion Criteria:

1. Smokers.
2. Pregnant and breast-feeding females.
3. Mentally retarded Patients.
4. Presence of hematologic disease.
5. Previous radiation, chemotherapy, or immunosuppressive treatments.
6. Diabetes mellitus, metabolic bone disease, ongoing treatment with bisphosphonates drugs, or pregnancy.
7. Patient with history of chronic sinus pathosis
8. Anticoagulant drugs, Endocarditis risk factors, renal and hepatic failure.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-26 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
histomorphometric analysis | 3 months
  After three months from sinus augmentation, a second surgery will be done for implant placement; during this procedure, a bone core biopsy will be harvested. The biopsy will be stained with mason stain for histomorphometric analysis. The aim is to measure the newly formed bone for three months.

IPD SHARING:
Plan to Share IPD: Undecided